CLINICAL TRIAL: NCT03894969
Title: Immunogenicity and Safety Study of GSK's Investigational Vaccine (GSK3277511A) When Administered in Healthy Smokers and Ex-smokers Following Receipt of Shingrix Vaccine
Brief Title: Study to Assess the Immunogenicity and Safety of GSK's Investigational Vaccine (GSK3277511A) When Given to Healthy Smokers and Ex-smokers After Administration of Shingrix Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 209538; 2018-002977-24 (EudraCT Number)
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Results first posted 2021-09-27 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Disorders
Keywords: Immunogenicity; Chronic obstructive pulmonary disease (COPD); Non-typeable Haemophilus influenza; Moraxella catarrhalis; Shingrix; Herpes Zoster; Adjuvanted vaccines; Safety
MeSH Terms: conditions — Respiration Disorders; Pulmonary Disease, Chronic Obstructive; Herpes Zoster | interventions — Acyl-Carrier Protein S-Malonyltransferase; Vaccines

STUDY DESIGN:
Masking Description: This is an open-label study. Blinding was not performed on the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Sh_NTHi-Mcat_1 Group (Experimental): Subjects enrolled in this group received 2 doses of GSK Biologicals' Shingrix vaccine at Day 1 and Day 61, and following a 1-month gap, subjects received 2 doses of GSK Biological's NTHi-Mcat investigational vaccine 2 months apart, at Day 91, and Day 151.
  Interventions: Biological: GSK's investigational non-typeable Haemophilus influenzae (NTHi) and Moraxella catarrhalis (Mcat) multi-antigen vaccine (GSK3277511A) adjuvanted with AS01E; Biological: Shingrix GSK's lyophilized formulation of the herpes zoster (HZ) vaccine (GSK1437173A)
- Sh_NTHi-Mcat_3 Group (Experimental): Subjects enrolled in this group received 2 doses of GSK Biologicals' Shingrix vaccine at Day 1 and Day 61 and, following a 3-month gap, subjects received 2 doses of GSK Biological's NTHi-Mcat investigational vaccine 2 months apart, at Day 151 and Day 211.
  Interventions: Biological: GSK's investigational non-typeable Haemophilus influenzae (NTHi) and Moraxella catarrhalis (Mcat) multi-antigen vaccine (GSK3277511A) adjuvanted with AS01E; Biological: Shingrix GSK's lyophilized formulation of the herpes zoster (HZ) vaccine (GSK1437173A)
- Sh_NTHi-Mcat_6 Group (Experimental): Subjects enrolled in this group received 2 doses of GSK Biologicals' Shingrix vaccine at Day 1 and Day 61 and, following a 6-month gap, subjects received 2 doses of GSK Biological's NTHi-Mcat investigational vaccine 2 months apart at Day 241 and Day 301.
  Interventions: Biological: GSK's investigational non-typeable Haemophilus influenzae (NTHi) and Moraxella catarrhalis (Mcat) multi-antigen vaccine (GSK3277511A) adjuvanted with AS01E; Biological: Shingrix GSK's lyophilized formulation of the herpes zoster (HZ) vaccine (GSK1437173A)
- NTHi-Mcat Group (Active Comparator): Subjects enrolled in this group received 2 doses of GSK Biological's NTHi-Mcat investigational vaccine 2 months apart, at Day 1 and Day 61.
  Interventions: Biological: GSK's investigational non-typeable Haemophilus influenzae (NTHi) and Moraxella catarrhalis (Mcat) multi-antigen vaccine (GSK3277511A) adjuvanted with AS01E
- Shingrix-Only Group (Experimental): Subjects belonging to this group were originally randomized to either Sh_NTHi-Mcat_1 Group, Sh_NTHi-Mcat_3 Group or Sh_NTHi-Mcat_6 Group, they received at least 1, maximum 2 doses of GSK Biologicals Shingrix vaccine at Day 1 and Day 61, but didnt receive any dose of NTHI Mcat investigational vaccine. Only safety data were collected for these subjects.
  Interventions: Biological: Shingrix GSK's lyophilized formulation of the herpes zoster (HZ) vaccine (GSK1437173A)

INTERVENTIONS:
Biological: GSK's investigational non-typeable Haemophilus influenzae (NTHi) and Moraxella catarrhalis (Mcat) multi-antigen vaccine (GSK3277511A) adjuvanted with AS01E — 2 doses of the investigational NTHi-Mcat vaccine will be administered 2 months apart to all subjects in all the groups. The vaccine will be given intramuscularly (IM) in the upper deltoid of non-dominant arm
  Arms: NTHi-Mcat Group; Sh_NTHi-Mcat_1 Group; Sh_NTHi-Mcat_3 Group; Sh_NTHi-Mcat_6 Group
Biological: Shingrix GSK's lyophilized formulation of the herpes zoster (HZ) vaccine (GSK1437173A) — 2 doses of the Shingrix vaccine will be administered at days 1 and 61 to all subjects in groups Sh_NTHi-Mcat_1, 3 and 6. The vaccine will be given intramuscularly (IM) in the upper deltoid of the non-dominant arm
  Arms: Sh_NTHi-Mcat_1 Group; Sh_NTHi-Mcat_3 Group; Sh_NTHi-Mcat_6 Group; Shingrix-Only Group

SUMMARY:
This study will provide information regarding the sequential administration of two vaccines adjuvanted with AS01.

The aim of this study is to understand immunogenicity and safety of NTHi-Mcat vaccine when administered sequentially after Shingrix vaccine and to compare to the immunogenicity of NTHi-Mcat vaccine administered alone. This study will also provide information regarding whether a specific time period is required between the administration of these two different vaccines containing the same adjuvant- AS01 components.

The population of this study will include healthy smokers and ex-smokers of 50 to 80 years of age which will be used as a proxy for the COPD population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* Written informed consent obtained from the subject prior to performance of any study specific procedure.
* A male or female between, and including, 50 years and 80 years of age at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Current or former smoker with a cigarette smoking history ≥10 pack-years.
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject: has practiced adequate contraception for 30 days prior to vaccination, and; has a negative pregnancy test on the day of vaccination, and; has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Medical conditions
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of potential immune-mediated disease (pIMD). Note: If the subject has any condition on the list of pIMDs specified in the protocol, they must be excluded unless the aetiology is clearly documented to be non-immune mediated.

The investigator will exercise his/her medical and scientific judgement in deciding whether other diseases have an autoimmune origin and thus meet the exclusion criteria.

* Diagnosis of COPD regardless of severity.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines. Additionally, consider allergic reactions to other material or equipment related to study participation (such as materials that may possibly contain latex -gloves, syringes, etc).
* Has significant disease (including significant psychological disorders), in the opinion of the investigator, likely to interfere with the study and/or likely to cause death within the study duration.
* History of or current condition preventing intramuscular injection as bleeding or coagulation disorder.
* Malignancies within previous 5 years (excluding non-melanoma skin cancer) or lymphoproliferative disorders.
* Prior/concomitant therapy
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines during the period starting 30 days before the first dose of study vaccine (Day -29 to Day 1), or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine administration, with the exception of non-MF59 adjuvanted influenza vaccines and pneumococcal vaccines which may be administered ≥15 days preceding or following any study vaccine dose.

Note: For M59 adjuvanted flu vaccine and for any vaccine containing novel adjuvant refer to exclusion criteria below.

* Planned administration/administration of a vaccine adjuvanted with the following adjuvants AS01, AS02, AS03, AS04 and MF59 in the period starting 6 months before the first dose of study vaccine, and ending at the second blood draw (i.e. approximately 1 month after the administration of the last dose of NTHi-Mcat vaccine). The following non-exhaustive list should be considered as criteria for exclusion: Prepandrix, Adjupanrix, Shingrix, Fendrix, Cervarix, FluAd, Chiromas, Gripguard.
* Previous vaccination with any vaccine containing NTHi and/or Mcat antigens
* Previous vaccination with Shingrix; (either registered product or participation in a previous vaccine study).
* Previous vaccination with HZ live-attenuated vaccine (ZVL)) (either registered product or participation in a previous vaccine study) within the 2 months of the first study visit (Day 1).
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 6 months prior to the first vaccine dose, and ending at the second blood draw. (i.e. approximately 1 month after the administration of the last dose of NTHi-Mcat vaccine). For corticosteroids, this will mean prednisone ≥5 mg/day (for adult subjects), or equivalent. Only topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the first dose of study vaccine or planned administration starting from Day 1 and ending at the second blood draw (i.e. approximately 1 month after the planned administration of the second dose of NTHi-Mcat vaccine).
* Prior/concurrent clinical study experience
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or medical device).
* Other exclusions:
* Pregnant or lactating female,
* Female planning to become pregnant or planning to discontinue contraceptive precautions,
* Current alcoholism and/or drug abuse,
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study
* Any study personnel or immediate dependents, family, or household member.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (4):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (3):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rennes
- Italy (2):
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Verona, Veneto
- GSK Investigational Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Galgani I, Poder A, Jogi R, Anttila VJ, Milleri S, Borobia AM, Launay O, Testa M, Casula D, Grassano L, Tasciotti A, Dozot M, Arora AK. Immunogenicity and safety of the non-typable Haemophilus influenzae-Moraxella catarrhalis (NTHi-Mcat) vaccine administered following the recombinant zoster vaccine versus administration alone: Results from a randomized, phase 2a, non-inferiority trial. Hum Vaccin Immunother. 2023 Dec 31;19(1):2187194. doi: 10.1080/21645515.2023.2187194. Epub 2023 Mar 28. PMID 36974988
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 542 participants were enrolled in the study, but only 541 received at least 1 dose of study treatment (i.e. Shingrix and/or NTHi Mcat vaccine).
Period: Overall Study
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group | Shingrix-Only Group
Started | 134 | 134 | 122 | 135 | 16
Completed | 129 | 129 | 118 | 128 | 2
Not Completed | 5 | 5 | 4 | 7 | 14
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 2
Not completed — Lost to Follow-up | 3 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 4 | 8
Not completed — Other | 0 | 0 | 0 | 0 | 3
Not completed — Unsolicited Non-Serious Advers Event | 0 | 0 | 0 | 2 | 1
Not completed — Solicited Adverse Event | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group | Shingrix-Only Group | Total
Number analyzed (Participants) | 134 | 134 | 122 | 135 | 16 | 541
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (7.0) | 60.9 (6.7) | 60.5 (7.1) | 60.0 (7.1) | 62.4 (5.5) | 60.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 66 | 58 | 65 | 7 | 259
  Male | 71 | 68 | 64 | 70 | 9 | 282
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 1 | 0 | 0 | 1 | 0 | 2
  Black Or African American | 0 | 1 | 0 | 1 | 0 | 2
  Not Reported | 0 | 0 | 0 | 0 | 1 | 1
  Other | 4 | 3 | 2 | 4 | 4 | 17
  White | 129 | 130 | 120 | 129 | 11 | 519

OUTCOME MEASURES:

1. Primary Outcome: Anti-Protein D (PD), Anti-Protein E (PE), Anti-type IV Pili Subunit (PilA) and Anti-ubiquitous Surface Protein A2 of Moraxella Catarrhalis (UspA2) Adjusted Geometric Mean Concentrations (GMCs), One-month Post Dose-2 of NTHi-Mcat Vaccine
Description: Antibody concentrations as measured by ELISA (Enzyme-linked immunosorbent assay) and expressed as adjusted (ANCOVA model) GMCs in ELISA units per milliliter (EU/mL). Cut-off value for the assay is 153, 16, 8 and 28 EU/mL for Anti-PD, Anti-PE, Anti-PilA and Anti-UspA2 antibodies respectively. The ANCOVA model includes study group, smoking status (current or former), age category (50-59, 60-69, 70-80 years of age) and center as factors and the antibody concentration before Dose 1 as covariate. As per protocol set (PPS) sample size was not met in Sh_NTHi_Mcat_3 and Sh_NTHi-Mcat_6 groups then timeframe was adapted as follows: At 1 month after dose 2 of NTHi-Mcat vaccine (Day 181 in Sh_NTHi-Mcat_1 group and Day 91 in NTHi-Mcat group)
Time Frame: At 1 month after dose 2 of NTHi-Mcat vaccine (Day 181, in Sh_NTHi-Mcat_1 group and Day 91 in NTHi-Mcat group)
Population: Analysis was performed on the per protocol set (PPS) which included all subjects who received full study treatment course to which they were randomized and had post-vaccination immunogenicity data minus subjects with protocol deviations that lead to exclusion.According to protocol,as PPS sample size for Sh_NTHI_Mcat_3 and Sh_NTHI_Mcat_6 Groups was not met,those were not part of the analysis. Shingrix-Only Group was not included in this analysis,as subjects didn't receive the NTHi MCAT vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Sh_NTHi-Mcat_1 Group | NTHi-Mcat Group
Number analyzed (Participants) | 118 | 124
EU/mL
  Anti-PD: number analyzed (Participants) | 118 | 123
  Anti-PD | 1402.804 [1139.194 to 1727.414] | 1489.531 [1203.846 to 1843.014]
  Anti-PE | 6234.827 [5053.049 to 7692.992] | 7032.52 [5666.105 to 8728.452]
  Anti-PilA: number analyzed (Participants) | 117 | 124
  Anti-PilA | 1244.373 [963.063 to 1607.854] | 1089.799 [840.246 to 1413.47]
  Anti-UspA2 | 1022.961 [894.403 to 1169.998] | 941.45 [820.993 to 1079.58]
Statistical Analysis 1: Comparison: Sh_NTHi-Mcat_1 Group; To demonstrate the non-inferiority (NI) of the humoral immune response 1 month after Dose 2 of GSK Biologicals' NTHi-Mcat investigational vaccine when administered 1 after Shingrix vaccine versus the humoral immune response 1 month after Dose 2 of GSKBiologicals' NTHi-Mcat investigational vaccine alone; Test type: Non-Inferiority — Non-inferiority is concluded if the lower limit of the two sided 95% CI for the GMC ratio for anti-PD is > 0.667. The anti-PD GMC ratio is presented in this test with its 95% CI; ANCOVA; ANCOVA model with treatment group, age category, smoking status and center as fixed effects and pre-Dose 1 log-concentration as a covariate; GMC ratio = 0.942, .95% CI 2-sided [0.765 to 1.159]
Statistical Analysis 2: Comparison: Sh_NTHi-Mcat_1 Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Non-inferiority is concluded if the lower limit of the two sided 95% CI for the GMC ratio for anti-PE is > 0.667. The anti-PE GMC ratio is presented in this test with its 95% CI; ANCOVA; [statistical method as in outcome 1, analysis 1]; GMC ratio = 0.887, .95% CI 2-sided [0.719 to 1.093]
Statistical Analysis 3: Comparison: Sh_NTHi-Mcat_1 Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Non-inferiority is concluded if the lower limit of the two sided 95% CI for the GMC ratio for anti-PilA is > 0.667. The anti-PilA GMC ratio is presented in this test with its 95% CI; ANCOVA; [statistical method as in outcome 1, analysis 1]; GMC ratio = 1.142, .95% CI 2-sided [0.884 to 1.474]
Statistical Analysis 4: Comparison: Sh_NTHi-Mcat_1 Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Non-inferiority is concluded if the lower limit of the two sided 95% CI for the GMC ratio for anti-UspA2 is > 0.667. The anti-UspA2 GMC ratio is presented in this test with its 95% CI; ANCOVA; [statistical method as in outcome 1, analysis 1]; GMC ratio = 1.087, .95% CI 2-sided [0.948 to 1.245]

2. Secondary Outcome: Anti-PD, Anti-PE, Anti-PilA, Anti-UspA2 Antibody Concentrations in Terms of GMCs, Before First NTHi-Mcat Vaccine
Description: GMCs and their 95% CI for each of the antibodies, as measured by ELISA, were calculated (the GMCs were computed by taking the Anti-log of the mean of the log concentration transformations)
Time Frame: Before the first dose of NTHi-Mcat vaccine (Day 91, Day 151 and Day 241 for Sh_NTHi-Mcat_1, Sh_NTHi-Mcat_3 and Sh_NTHi-Mcat_6 group, respectively, and Day 1 for NTHi-Mcat group)
Population: Analysis was performed on the PPS which included all subjects who received full study treatment course to which they were randomized and had post-vaccination immunogenicity data minus subjects with protocol deviations that lead to exclusion. Subjects from the Shingrix-Only Group were not included in this analysis, as they didn't receive the NTHi MCAT vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group
Number analyzed (Participants) | 118 | 96 | 73 | 124
EU/mL
  Anti-PD: number analyzed (Participants) | 118 | 95 | 73 | 124
  Anti-PD | 94.7 [86.2 to 104.1] | 105.1 [89.8 to 123] | 95.6 [84.5 to 108.3] | 105.3 [93.4 to 118.6]
  Anti-PE: number analyzed (Participants) | 118 | 96 | 73 | 123
  Anti-PE | 22 [18 to 26.9] | 21.2 [17.6 to 25.4] | 18.6 [14.3 to 24.2] | 23.9 [19.8 to 28.9]
  Anti-PilA | 7.8 [6.6 to 9.3] | 10.5 [8.2 to 13.5] | 9.7 [7.5 to 12.6] | 9.1 [7.5 to 11]
  Anti-UspA2 | 352.4 [292.5 to 424.7] | 343 [286.3 to 411] | 440.3 [343.5 to 564.5] | 521.4 [441 to 616.3]

3. Secondary Outcome: Anti-PD, Anti-PE, Anti-PilA, Anti-UspA2 Antibody Concentrations in Terms of GMCs, One-month Post Dose-2 of NTHi-Mcat Vaccine
Description: GMCs and their 95% CI for each of the antibodies, as measured by ELISA, were calculated (the GMCs were computed by taking the Anti-log of the mean of the log concentration transformations) before the first dose of NTHi-Mcat vaccine
Time Frame: At one month after the second dose of NTHi-Mcat vaccine (Day 181, 241, 331 in the Sh_NTHi-Mcat_1, Sh_NTHi-Mcat_3 and Sh_NTHi-Mcat_6 group, respectively, and Day 91 in the NTHi-Mcat group)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group
Number analyzed (Participants) | 118 | 96 | 73 | 124
EU/mL
  Anti-PD: number analyzed (Participants) | 118 | 96 | 73 | 123
  Anti-PD | 1496.7 [1272.7 to 1760.1] | 1504 [1209.9 to 1869.6] | 1539 [1277.3 to 1854.2] | 1683.5 [1434.5 to 1975.5]
  Anti-PE | 5911.8 [5121.3 to 6824.3] | 5920.8 [4868.4 to 7200.8] | 6048.5 [4943.3 to 7400.8] | 6562.4 [5660.9 to 7607.5]
  Anti-PilA: number analyzed (Participants) | 117 | 96 | 73 | 124
  Anti-PilA | 1089.3 [910.3 to 1303.4] | 1030.6 [839.4 to 1265.3] | 1114.7 [864.9 to 1436.6] | 999.3 [830.3 to 1202.7]
  Anti-UspA2 | 926.8 [796.6 to 1078.4] | 942.2 [819.6 to 1083.2] | 1289.2 [1062.5 to 1564.5] | 1066.4 [946.6 to 1201.4]

4. Secondary Outcome: Percentage of Seropositive Subjects for Anti-PD, Anti-PE, Anti-PilA, Anti-UspA2 Antibodies Before First NTHi-Mcat Vaccine
Description: A seropositive subject is defined as a subject whose Anti-PD, Anti-PE, Anti-PilA and Anti-UspA2 antibody concentrations are greater than or equal to the assay cut-off value. Seropositivity rates with 95% CI is defined using the assay lower limit of quantification (LLOQ). Cut-off value for the assay is 153, 16, 8 and 28 EU/mL for Anti-PD, Anti-PE, Anti-PilA and Anti-UspA2 antibodies respectively
Time Frame: Before the first dose of NTHi-Mcat vaccine (Day 91, Day 151 and Day 241 in the Sh_NTHi-Mcat_1, Sh_NTHi-Mcat_3 and Sh_NTHi-Mcat_6 group, respectively, and Day 1 in the NTHi-Mcat group)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group
Number analyzed (Participants) | 118 | 96 | 73 | 124
Percentage of subjects
  Anti-PD: number analyzed (Participants) | 118 | 95 | 73 | 124
  Anti-PD | 16.9 [10.7 to 25] | 20 [12.5 to 29.5] | 19.2 [10.9 to 30.1] | 21.8 [14.9 to 30.1]
  Anti-PE: number analyzed (Participants) | 118 | 96 | 73 | 123
  Anti-PE | 57.6 [48.2 to 66.7] | 63.5 [53.1 to 73.1] | 50.7 [38.7 to 62.6] | 61.8 [52.6 to 70.4]
  Anti-PilA | 38.1 [29.4 to 47.5] | 49 [38.6 to 59.4] | 47.9 [36.1 to 60] | 43.5 [34.7 to 52.7]
  Anti-UspA2 | 100 [96.9 to 100] | 100 [96.2 to 100] | 100 [95.1 to 100] | 100 [97.1 to 100]

5. Secondary Outcome: Percentage of Subjects Seropositive for Anti-PD, Anti-PE, Anti-PilA, Anti-UspA2 Antibodies, One-month Post Dose-2 of NTHi-Mcat Vaccine
Description: A seropositive subject is defined as a subject whose Anti-PD, Anti-PE, Anti-PilA and Anti-UspA2 antibody concentrations are greater than or equal to the assay cut-off value. Seropositivity rates with 95% CI are defined using the assay (LLOQ). Cut-off value for the assay is 153, 16, 8 and 28 EU/mL for Anti-PD, Anti-PE, Anti-PilA and Anti-UspA2 antibodies respectively
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group
Number analyzed (Participants) | 118 | 96 | 73 | 124
Percentage of subjects
  Anti-PD: number analyzed (Participants) | 118 | 96 | 73 | 123
  Anti-PD | 99.2 [95.4 to 100] | 97.9 [92.7 to 99.7] | 100 [95.1 to 100] | 100 [97 to 100]
  Anti-PE | 100 [96.9 to 100] | 100 [96.2 to 100] | 100 [95.1 to 100] | 100 [97.1 to 100]
  Anti-PilA: number analyzed (Participants) | 117 | 96 | 73 | 124
  Anti-PilA | 100 [96.9 to 100] | 100 [96.2 to 100] | 100 [95.1 to 100] | 100 [97.1 to 100]
  Anti-UspA2 | 100 [96.9 to 100] | 100 [96.2 to 100] | 100 [95.1 to 100] | 100 [97.1 to 100]

6. Secondary Outcome: Frequency of Specific Cluster of Differentiation 4 (CD4+) T-cells Against NTHi and Mcat Antigens for Evaluation of Cell-mediated Immune (CMI) Response, Before First Dose of NTHi-Mcat Vaccine
Description: Frequency of specific CD4+ T-cells was measured by flow cytometry intracellular cytokine staining (ICS) expressing at least 2 different markers among CD40 Ligand (CD40L), interleukin (IL)-2, IL-13, IL-17, tumour necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ), upon in vitro stimulation
Time Frame: as for outcome 4
Population: Analysis was performed on Cell-Mediated immune (CMI) sub-cohort, which included approximately 60 subjects (15/each group), for which an additional blood sample was taken at each pre-defined timepoint (sub-cohort selected from sites able to process the blood samples according to GSK procedures for peripheral blood mononuclear cell preparation). Subjects from the Shingrix-Only Group were not included in this analysis, as they didn't receive the NTHi MCAT vaccine.
Measure: Mean (Standard Deviation); unit: CD4+ T cells/million cells
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group
Number analyzed (Participants) | 10 | 12 | 3 | 13
CD4+ T cells/million cells
  M catarrhalis.UspA2 - CD4+ T-cells | 112.945 (153.903) | 101.739 (94.932) | 81.578 (90.919) | 92.685 (99.661)
  NTHi.PD - CD4+ T-cells | 89.456 (68.929) | 59.522 (82.06) | 36.439 (57.347) | 96.893 (74.87)
  NTHi.PE - CD4+ T-cells | 79.838 (58.999) | 46.112 (63.007) | 69.546 (97.09) | 80.717 (119.316)
  NTHi.PilA - CD4+ T-cells | 61.627 (53.613) | 42.438 (55.575) | 60.139 (51.37) | 105.558 (97.618)

7. Secondary Outcome: Frequency of CD4+ T-cells Against NTHi and Mcat Antigens for Evaluation of CMI Response, at One-month Post Dose 2 of NTHi-Mcat Vaccine
Description: Frequency of specific CD4+ T-cells was measured by flow cytometry ICS expressing at least 2 different markers among CD40L, IL-2, IL-13, IL-17, TNF-α and IFN-γ, upon in vitro stimulation
Time Frame: At one month after second dose of NTHi-Mcat vaccine (Day 181, Day 241 and Day 331 in the Sh_NTHi-Mcat_1, Sh_NTHi-Mcat_3 and Sh_NTHi-Mcat_6 group, respectively, and Day 91 in the NTHi-Mcat group)
Population: Analysis was performed on CMI sub-cohort, which included approximately 60 subjects (15/each group), for which an additional blood sample was taken at each pre-defined time point (sub-cohort selected from sites able to process the blood samples according to GSK procedures for peripheral blood mononuclear cell preparation). Subjects from the Shingrix-Only Group were not included in this analysis, as they didn't receive the NTHi MCAT vaccine.
Measure: Mean (Standard Deviation); unit: CD4+ T cells/million cells
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group
Number analyzed (Participants) | 10 | 11 | 3 | 13
CD4+ T cells/million cells
  M catarrhalis.UspA2 - CD4+ T-cells | 721.851 (457.94) | 619.68 (392.133) | 1001.839 (144.057) | 735.177 (471.515)
  NTHi.PD - CD4+ T-cells | 632.849 (323.731) | 527.26 (281.827) | 1570.631 (1064.327) | 742.666 (527.567)
  NTHi.PE - CD4+ T-cells | 565.964 (411.715) | 581.338 (520.594) | 888.057 (154.524) | 1155.341 (699.841)
  NTHi.PilA - CD4+ T-cells | 332.43 (273.215) | 318.46 (195.527) | 333.501 (121.712) | 388.282 (207.434)

8. Secondary Outcome: Percentage of Subjects With Reported Solicited Local Adverse Event (AE)
Description: The percentage of subjects with at least one local solicited AE, regardless of intensity, during the 7-day follow-up period after each NTHi-Mcat vaccine dose, are reported by study group. Assessed local symptoms were pain, redness and swelling. Any local injection site redness/swelling is scored as follows: diameter >=20 milli-meters
Time Frame: During the 7-day follow-up period (i.e. day of vaccination and 6 subsequent days) after Dose 1 and after Dose 2 of NTHi-Mcat vaccine
Population: Analysis was performed on the Solicited safety set (SSS) which included all subjects who received at least 1 dose of the study treatment and who have solicited safety data
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group
Number analyzed (Participants) | 134 | 133 | 118 | 135
Percentage of subjects
  Erythema (mm), Dose 1 | 6 [2.6 to 11.4] | 15 [9.4 to 22.3] | 11 [6 to 18.1] | 12.6 [7.5 to 19.4]
  Erythema (mm), Dose 2: number analyzed (Participants) | 133 | 131 | 117 | 127
  Erythema (mm), Dose 2 | 12.8 [7.6 to 19.7] | 13.7 [8.4 to 20.8] | 17.9 [11.5 to 26.1] | 11.8 [6.8 to 18.7]
  Pain, Dose 1 | 59.7 [50.9 to 68.1] | 69.2 [60.6 to 76.9] | 61 [51.6 to 69.9] | 63.7 [55 to 71.8]
  Pain, Dose 2: number analyzed (Participants) | 133 | 131 | 117 | 127
  Pain, Dose 2 | 69.9 [61.4 to 77.6] | 76.3 [68.1 to 83.3] | 72.6 [63.6 to 80.5] | 75.6 [67.2 to 82.8]
  Swelling (mm), Dose 1 | 3.7 [1.2 to 8.5] | 10.5 [5.9 to 17] | 5.9 [2.4 to 11.8] | 5.2 [2.1 to 10.4]
  Swelling (mm), Dose 2: number analyzed (Participants) | 133 | 131 | 117 | 127
  Swelling (mm), Dose 2 | 7.5 [3.7 to 13.4] | 8.4 [4.3 to 14.5] | 6.8 [3 to 13] | 7.9 [3.8 to 14]

9. Secondary Outcome: Percentage of Subjects With Reported Solicited General AE
Description: The percentage of subjects with at least one general solicited AE, regardless of intensity, during the 7-day follow-up period after each NTHi-Mcat vaccine dose, are reported by study group. Assessed solicited general symptoms were Fatigue, Gastrointestinal symptoms (nausea, vomiting, diarrhoea and/or abdominal pain), Headache, Myalgia, Chills and Fever (oral cavity or axillary route - temperature equal or higher than [>=] 37.5 degrees Celsius [°C])
Time Frame: as for outcome 8
Population: Analysis was performed on the SSS which included all subjects who received at least 1 dose of the study treatment and who have solicited safety data
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group
Number analyzed (Participants) | 134 | 133 | 118 | 135
Percentage of subjects
  Chills, Dose 1 | 11.9 [7 to 18.7] | 12 [7 to 18.8] | 16.9 [10.7 to 25] | 7.4 [3.6 to 13.2]
  Chills, Dose 2: number analyzed (Participants) | 133 | 131 | 117 | 127
  Chills, Dose 2 | 25.6 [18.4 to 33.8] | 26 [18.7 to 34.3] | 22.2 [15.1 to 30.8] | 16.5 [10.5 to 24.2]
  Fatigue, Dose 1 | 26.1 [18.9 to 34.4] | 38.3 [30.1 to 47.2] | 39 [30.1 to 48.4] | 34.1 [26.1 to 42.7]
  Fatigue, Dose 2: number analyzed (Participants) | 133 | 131 | 117 | 127
  Fatigue, Dose 2 | 39.1 [30.8 to 47.9] | 48.1 [39.3 to 57] | 43.6 [34.4 to 53.1] | 37.8 [29.3 to 46.8]
  Fever (C), Dose 1 | 1.5 [0.2 to 5.3] | 1.5 [0.2 to 5.3] | 2.5 [0.5 to 7.3] | 3 [0.8 to 7.4]
  Fever (C), Dose 2: number analyzed (Participants) | 133 | 131 | 117 | 127
  Fever (C), Dose 2 | 11.3 [6.5 to 17.9] | 8.4 [4.3 to 14.5] | 8.5 [4.2 to 15.2] | 8.7 [4.4 to 15]
  Gastrointestinal symptoms, Dose 1 | 13.4 [8.2 to 20.4] | 13.5 [8.2 to 20.5] | 16.1 [10 to 24] | 13.3 [8.1 to 20.3]
  Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 133 | 131 | 117 | 127
  Gastrointestinal symptoms, Dose 2 | 15.8 [10 to 23.1] | 15.3 [9.6 to 22.6] | 12.8 [7.4 to 20.3] | 9.4 [5 to 15.9]
  Headache, Dose 1 | 20.9 [14.4 to 28.8] | 26.3 [19.1 to 34.7] | 22.9 [15.7 to 31.5] | 18.5 [12.4 to 26.1]
  Headache, Dose 2: number analyzed (Participants) | 133 | 131 | 117 | 127
  Headache, Dose 2 | 32.3 [24.5 to 41] | 38.2 [29.8 to 47.1] | 23.9 [16.5 to 32.7] | 22 [15.2 to 30.3]
  Myalgia, Dose 1 | 20.1 [13.7 to 27.9] | 23.3 [16.4 to 31.4] | 25.4 [17.9 to 34.3] | 27.4 [20.1 to 35.7]
  Myalgia, Dose 2: number analyzed (Participants) | 133 | 131 | 117 | 127
  Myalgia, Dose 2 | 33.1 [25.2 to 41.8] | 37.4 [29.1 to 46.3] | 36.8 [28 to 46.2] | 37.8 [29.3 to 46.8]

10. Secondary Outcome: Percentage of Subjects With Any Unsolicited AE
Description: An unsolicited adverse event is an adverse event that was not solicited using a Subject Diary and that was spontaneously communicated by a subject who has signed the informed consent. The percentage of subjects with at least one unsolicited AE, regardless of intensity or relationship to vaccination, during the 30-day follow-up period after any NTHi-Mcat vaccine dose are reported for each group. Any solicited symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event
Time Frame: During the 30-day follow-up period (i.e. day of vaccination and 29 subsequent days) after Dose 1 and after Dose 2 of NTHi-Mcat vaccine
Population: Analysis was performed on the Unsolicited safety set which included all subjects who receive at least 1 dose of the study treatment and who have unsolicited safety data
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group
Number analyzed (Participants) | 134 | 134 | 122 | 135
Percentage of subjects
  Dose 1 | 13.4 [8.2 to 20.4] | 14.9 [9.4 to 22.1] | 11.5 [6.4 to 18.5] | 18.5 [12.4 to 26.1]
  Dose 2: number analyzed (Participants) | 133 | 131 | 118 | 129
  Dose 2 | 15 [9.4 to 22.3] | 15.3 [9.6 to 22.6] | 8.5 [4.1 to 15] | 10.9 [6.1 to 17.5]

11. Secondary Outcome: Percentage of Subjects With Any Serious Adverse Event (SAE) During Epoch 001
Description: The percentage of subjects with at least one SAE, regardless of intensity or relationship to vaccination, from Day 1 up to and including Day 331, were reported for each group An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject or was a congenital anomaly/birth defect in the offspring of a study subject. AE(s) considered as SAE(s) also include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, as per the medical or scientific judgement of the physician
Time Frame: From Day 1 up to and including Day 331 (Epoch 001)
Population: Analysis was performed on the Exposed Set (ES) which included all subjects who received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group | Shingrix-Only Group
Number analyzed (Participants) | 134 | 134 | 122 | 135 | 16
Percentage of subjects | 4.5 [1.7 to 9.5] | 3.7 [1.2 to 8.5] | 2.5 [0.5 to 7] | 1.5 [0.2 to 5.2] | 6.3 [0.2 to 30.2]

12. Secondary Outcome: Percentage of Subjects With Any Potential Immune-mediated Diseases (pIMD's) During Epoch 001
Description: pIMD's are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Day 1 up to and including Day 331 (Epoch 001)
Population: Analysis was performed on the ES which included all subjects who received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group | Shingrix-Only Group
Number analyzed (Participants) | 134 | 134 | 122 | 135 | 16
Percentage of subjects | 0 [0 to 2.7] | 1.5 [0.2 to 5.3] | 0.8 [0 to 4.5] | 0 [0 to 2.7] | 12.5 [1.6 to 38.3]

13. Secondary Outcome: Percentage of Subjects With Any SAE During Epoch 002
Description: The percentage of subjects with at least one SAE, regardless of intensity or relationship to vaccination, from Day 332 up to and including Day 661, are reported for each group. An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, requires hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject or was a congenital anomaly/birth defect in the offspring of a study subject. AE(s) considered as SAE(s) also include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, as per the medical or scientific judgement of the physician.
Time Frame: From Day 332 up to and including Day 661 (Epoch 002)
Population: Analysis was performed on the ES which included all subjects who received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Shingrix-Only Group: Subjects enrolled in this group received at least 1, maximum 2 doses of GSK Biologicals' Shingrix vaccine at Day 1 and Day 61, but didn't receive any dose of NTHI Mcat investigational vaccine.
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group | Shingrix-Only Group
Number analyzed (Participants) | 134 | 134 | 122 | 135 | 16
Percentage of subjects | 3.0 [0.8 to 7.5] | 4.5 [1.7 to 9.5] | 3.3 [0.9 to 8.2] | 2.2 [0.5 to 6.4] | 0.0 [0.0 to 20.6]

14. Secondary Outcome: Percentage of Subjects With Any pIMD's During Epoch 002
Description: as for outcome 12
Time Frame: From Day 332 up to and including Day 661 (Epoch 002)
Population: Analysis was performed on the ES which included all subjects who received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group | Shingrix-Only Group
Number analyzed (Participants) | 134 | 134 | 122 | 135 | 16
Percentage of subjects | 0.7 [0.0 to 4.1] | 0.7 [0.0 to 4.1] | 0.0 [0.0 to 3.0] | 0.0 [0.0 to 2.7] | 0.0 [0.0 to 20.6]

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected during the 7-day follow-up period and unsolicited adverse events during the 30-day follow-up period. Serious adverse events were collected from Day 1 up to Day 661.
Description: Other Adverse events were not collected for Shingrix-Only Group.
Arm/Group | Sh_NTHi-Mcat_1 Group | Sh_NTHi-Mcat_3 Group | Sh_NTHi-Mcat_6 Group | NTHi-Mcat Group | Shingrix-Only Group
All-Cause Mortality (participants affected / at risk) | 0/134 | 1/134 | 0/122 | 0/135 | 0/16
Serious Adverse Events (participants affected / at risk) | 9/134 | 11/134 | 6/122 | 5/135 | 1/16
Other Adverse Events (participants affected / at risk) | 118/134 | 125/134 | 107/122 | 125/135 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sh_NTHi-Mcat_1 Group (N=134) | Sh_NTHi-Mcat_3 Group (N=134) | Sh_NTHi-Mcat_6 Group (N=122) | NTHi-Mcat Group (N=135) | Shingrix-Only Group (N=16)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sh_NTHi-Mcat_1 Group (N=134) | Sh_NTHi-Mcat_3 Group (N=134) | Sh_NTHi-Mcat_6 Group (N=122) | NTHi-Mcat Group (N=135) | Shingrix-Only Group (N=0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | NA
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | NA
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | NA
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 34 (39) | 32 (38) | 26 (34) | 26 (30) | NA
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | NA
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | NA
Chest discomfort (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | NA
Chills (General disorders) | 40 (50) | 41 (50) | 40 (47) | 26 (31) | NA
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Fatigue (General disorders) | 63 (88) | 78 (114) | 68 (99) | 65 (95) | NA
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Hangover (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA
Injection site erythema (General disorders) | 21 (25) | 27 (38) | 28 (34) | 24 (32) | NA
Injection site movement impairment (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Injection site pain (General disorders) | 105 (173) | 112 (192) | 98 (157) | 112 (182) | NA
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Injection site swelling (General disorders) | 12 (15) | 19 (25) | 13 (15) | 15 (17) | NA
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | NA
Pyrexia (General disorders) | 16 (17) | 12 (13) | 13 (13) | 14 (15) | NA
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Bronchitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | NA
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | NA
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | NA
Schistosomiasis cutaneous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | NA
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | NA
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | NA
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | NA
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | NA
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | NA
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 48 (73) | 64 (80) | 56 (76) | 67 (87) | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Headache (Nervous system disorders) | 56 (78) | 66 (92) | 44 (59) | 42 (56) | NA
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | NA
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | NA
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Dental implantation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT03894969/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03894969/SAP_001.pdf